CLINICAL TRIAL: NCT02297126
Title: A Prospective Randomized Trial to Assess Cost and Clinical Outcomes of a Clinical Pharmacogenomic Program at Eskenazi Hospital
Brief Title: A Prospective Trial to Assess Cost and Clinical Outcomes of a Clinical Pharmacogenomic Program
Acronym: INGenious
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Principal Investigator, Todd Skaar, PhD, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1401206188; U01HG007762-01 (NIH)
Record Dates: First submitted 2014-11-05; First posted 2014-11-21 (Estimated); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Adverse Drug Reaction
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Arm (No Intervention): 4,000 patients receiving a new prescription for targeted medication(s) randomized into the control arm receive standard care (no intervention affecting drug selection, dosage, dosage form, frequency and duration of therapy). Healthcare costs and adverse events data collected and analyzed for 12 months from time of entry into study. List of targeted medications: codeine, amitriptyline, aripiprazole, atazanavir, atomoxetine, azathioprine, citalopram, clopidogrel, cyclophosphamide, doxepin, efavirenz, escitalopram, esomeprazole, fluconazole, simvastatin, fluorouracil, phenytoin, quetiapine, glyburide, lansoprazole, mercaptopurine, methadone, methotrexate, nortriptyline, omeprazole, pantoprazole, rasburicase, tacrolimus, thioguanine, tramadol, venlafaxine, voriconazole and warfarin
- Pharmacogenetic Intervention Arm (Experimental): 2,000 patients receiving new prescription for targeted medication(s) identified in the control arm will be randomized to the intervention arm, consented and a tests will be performed from a blood sample. The treating physicians will be provided with the pharmacogenetic information and will determine if intervention is appropriate. Physician may elect to stay the course of therapy or alter drug selection, dosage, dosage form, frequency or duration of therapy based on the pharmacogenetic test results and input from clinical pharmacology consultations (if requested). Patients in the intervention arm will have their overall healthcare costs and clinical outcomes (specifically adverse events) followed and analyzed for a 1 year period from the time that they are entered into the study
  Interventions: Other: Pharmacogenetic Intervention Arm (pharmacogenetic testing)

INTERVENTIONS:
Other: Pharmacogenetic Intervention Arm (pharmacogenetic testing) — In the design of this trial, pharmacogenetic testing will be triggered by the incident prescription of one or more of the targeted medications listed in the control arm. The pharmacogenetic array to be used incorporates 51 genetic variants for the following 16 genes/transporters: ATP-binding cassette sub-family C member 2, ATP-binding cassette, sub-family C, member 4, Cytochrome P450 2B6, Cytochrome P450 2C19, Cytochrome P450 2C9, Cytochrome P450 2D6, Cytochrome P450 3A4/3A5, Cytochrome P450 4F2, Dihydropyrimidine dehydrogenase, Glucose-6-Phosphate Dehydrogenase, Human Leukocyte antigen-B, I interleukin-28B, Inosine Triphosphatase, Solute Carrier Organic Anion Transporter Family, Member 1B, Thiopurine methyltransferase and V vitamin K epoxide reductase complex, subunit 1.
  Arms: Pharmacogenetic Intervention Arm

SUMMARY:
The INGenious trial will prospectively enroll a total of 6,000 patients, with 2,000 patients assigned to a pharmacogenetic testing arm and 4,000 to a control arm who will be followed, but not tested. It is randomized between an intervention arm and one that receives no intervention in order that the genotyped group can be compared with one in which undisturbed, routine clinical care is carried out in patients taking the same drugs. Both arms will be followed for a year after being prescribed a targeted medication. Patients randomized into the intervention arm that are prescribed one or more of the 24 targeted index medication will receive pharmacogenomic testing using a custom micro-array measuring 51 Single nucleotide polymorphisms in 16 genes. The study is being conducted by the Indiana University School of Medicine and the Indiana University Institute of Personalized Medicine in collaboration with the Eskenazi and Indiana University Health Systems and will evaluate the economic and clinical outcomes associated with embedding a pharmacogenomics program in a system that serves as the primary health care safety-net in Indianapolis, Indiana. By successfully implementing a pharmacogenomics program and integrating it with the Electronic Health Record and Clinical Decision Support system, physicians will be able to optimize patient care by delivering tailored therapeutic decisions based on the patient's individual genetics.

DETAILED DESCRIPTION:
Indiana University School of Medicine and the Indiana University Institute of Personalized Medicine in collaboration with the Eskenazi Health and IUH Systems will be conducting a NIH funded randomized trial beginning in 2014. The study will evaluate the economic and clinical outcomes of associated with embedding a pharmacogenomics program in a system that serves as a health care safety-net in Indianapolis, Indiana, and handles over 1.2 million outpatient visits a year at its hospital and network of 10 community health centers. There are over 990,000 outpatient visits and 15,000 adult admissions annually, and the payor mix includes 45% uninsured, 26% Medicaid and 18% Medicare patients. This health care system has more than 40 years of experience in digital medical record implementation and a proven track record of innovation in medical informatics that is based in the Regenstrief Institute.

The goal of Personalized Medicine (PM) is to implement advances in biomarker pharmacology, molecular diagnostics and genomics to improve the health of patients afflicted by a wide range of medical conditions. Dramatic advances in genomics have identified numerous disease/therapeutic associations now placing this goal within sight. For the full benefits of personalized genomic medicine to be realized, it is now critical that progress made on a small scale be extended. The fruits of outstanding scientific discovery are often enjoyed by a small number of academic medical centers but are not scalable, and therefore not available to the masses of patients found in larger health care systems. In addition, such advances often bypass underserved populations, resulting significant inequalities of care.

Study Aims:

Aim 1: To test the hypothesis that a Clinical Laboratory Improvement Amendment certified genotyping targeted at 24 widely used drugs is associated with significant reductions in hospital and outpatient economic costs incurred over 1 year.

Aim2: To test whether pharmacogenetic testing is associated with significant improvements in clinical outcomes over 1 year.

The INGENIOUS trial will enroll a total of 6,000 patients, with 2,000 patients assigned to a pharmacogenetic testing arm and 4,000 to a control arm who will be followed, but not tested. The study is prospective since practice patterns change, and retrospective designs cannot be used to assess the impact of a prospective change. It is randomized between an intervention arm and one that receives no intervention in order that a genotyped group can be compared with one in which undisturbed, routine clinical care is carried out in patients taking the same drugs. Both arms will be followed for a year. Subjects will be enrolled starting at 6 months into the funding period, and investigators will enroll subjects for a total of 2 years, so that the last person enrolled will be at 2.5 years, and follow up will be completed at 3.5 years, allowing 6 months for analysis at the end of the study. A pharmacogenetic test, involving 51 Single nucleotide polymorphisms in 16 genes will be carried out at the beginning of the study in patients in the testing arm upon prompting by an index medication: one of 24 selected as being supported by validated guidelines.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if they are prescribed one of the 27 index medications for the first time, defined as there being no recorded prescription in the Eskenazi, Indiana University Health or Indiana Patient Care (INPC) system over the past year. The inclusion criteria that will be adhered to will be:

1. Able and willing consent to participation in the trial;
2. Adults aged 18 and over;
3. Receiving care at Eskenazi Health or Indiana University Health Systems for 1 year or more;
4. Prescribed an index medication.
5. No documented prescription of the index medication for the past year.
6. The study limit of enrollment (500) for that medication has not been reached
7. A single tube of whole blood can be obtained, and
8. Able to follow study procedures. -

Exclusion Criteria:

No subject will be excluded from the study on the basis of ethnicity or race. We will include all minorities.

Patients will be excluded if they:

1. Cannot or do not consent to participate;
2. are unable to provide 5cc of whole blood, or it cannot be obtained;
3. if they are an employee or student under the supervision of any of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4465 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Financial impact on the total cost of patient care resulting from implementation of a Pharmacogenetics testing program within a safety-net and Academic healthcare system | Study enrollment period of 2.5 years with individual patient data collection period of 12 month after one of more targeted medication is prescribed
  Analysis of cost of care (measured in U.S. dollars) data from the Eskenazi and Indiana University Health electronic medical records and billing systems for patients in the study. Charge data collected from monthly Eskenazi and IU Health System reports generated for the state hospital association. Categories of inpatient and outpatient charges include costs for medications, facility, laboratory, treatment, professional, and other sources. Data will be collected for each patient in the control and intervention arm beginning the day that the treating physician prescribes one or more targeted medication and will continue to be collected for 12 calendar months. Study enrollment period 2.5 years

SECONDARY OUTCOMES:
Impact of implementing a Pharmacogenetics program on Clinical Outcomes (incidence and severity of adverse events, frequency of healthcare visits, length of hospital stay, and readmissions) within a safety-net and Academic healthcare system | Study enrollment period of 2.5 years with individual patient data collection period of 12 month after one of more targeted medication is prescribed
  For each patient in the study, investigators from the Regenstrief Institute will collect 12 months of data from the Eskenazi and IUH electronic medical records and informatics systems beginning when one or more targeted medications are prescribed. Outcome measures include: number of patient admissions, readmissions, number of emergency department visits, number of clinic visits and returns to clinic. Data collected includes reported adverse drug reactions related to the targeted medications (utilizing text in the physician notes section of the medical record and records entered using International Classification of Diseases coding convention
Impact of implementing a Pharmacogenetics program on prescribing patterns within a safety-net healthcare system | Study enrollment period of 2.5 years with individual patient data collection period of 12 month after one of more targeted medication is prescribed
  Prescribing data will be collected for each patient in the control and intervention arm beginning the day that the treating physician prescribes one or more targeted medication and will continue to be collected for 12 calendar months. Study enrollment period 2.5 years. Medication possession ratio for index medications used to determine whether a change in drug regimen was implemented for the intervention versus the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Dexter, MD, Principal Investigator — Indiana University School of Medicine, Regenstrief Institute, Eskenazi Health; Todd Skaar, PhD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Eskenazi Health System, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy KD, Decker BS, Carpenter JS, Flockhart DA, Dexter PR, Desta Z, Skaar TC. Prerequisites to implementing a pharmacogenomics program in a large health-care system. Clin Pharmacol Ther. 2014 Sep;96(3):307-9. doi: 10.1038/clpt.2014.101. Epub 2014 May 7. PMID 24807457
- [Derived] Fulton CR, Zang Y, Desta Z, Rosenman MB, Holmes AM, Decker BS, Zhang Y, T Callaghan J, Pratt VM, Levy KD, Gufford BT, Dexter PR, Skaar TC, Eadon MT. Drug-gene and drug-drug interactions associated with tramadol and codeine therapy in the INGENIOUS trial. Pharmacogenomics. 2019 Apr;20(6):397-408. doi: 10.2217/pgs-2018-0205. Epub 2019 Feb 20. PMID 30784356